CLINICAL TRIAL: NCT05274633
Title: Real Life Use of Ravulizumab in Italian Patients With Paroxysmal Nocturnal Hemoglobinuria a Multicenter Observational Retrospective and Prospective Cohort Study.
Brief Title: Real Life Use of Ravulizumab in Italian Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMRAV601IT
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PIGA Gene; Complement-inhibitor Protein; CD55; CD59; Efficacy; Safety; Patient Registry
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With PNH: Data will be collected on participants who were already treated with eculizumab for at least 26 weeks and who started ravulizumab treatment as per clinical practice.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Participants will be observed for 52 weeks after the start of ravulizumab.
  Other Names: Ultomiris

SUMMARY:
This study will collect clinical response data on participants who were already treated with eculizumab for at least 26 weeks and who started ravulizumab treatment as a specific therapeutic strategy as per ordinary clinical practice.

DETAILED DESCRIPTION:
This study is an Italian multi-center, observational (non-interventional), cohort study composed of both retrospective and prospective observation periods on the same Paroxysmal Nocturnal Hemoglobinuria (PNH) participants. After the First Participant In from different Italian study centers, participants will be consecutively enrolled for 9 months and they will be observed for 52 weeks after the start of ravulizumab.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of 10 kilogram or above
* Hemolysis with clinical symptom(s) indicative of high disease activity
* Documented diagnoses of PNH confirmed by high-sensitivity flow cytometry evaluation of red blood cells and white blood cells with granulocyte or monocyte clone size of ≥ 5%
* Clinically stable after having been treated with eculizumab for at least the past 6 months
* Participant already assigned to ravulizumab treatment as a specific therapeutic strategy within the current routine clinical practice (this decision has to be made independently and before the enrolment of the participant in the study)
* Vaccinated against Neisseria meningitidis (according to Summary of Product Characteristics) < 3 years before dosing or at least 2 weeks prior to initiating ravulizumab unless the risk of delaying ravulizumab therapy outweighs the risk of developing a meningococcal infection
* Signed written informed and privacy consent prior to study participation

Exclusion Criteria:

* History of hematopoietic stem cell transplantation (evaluated at baseline)
* Known pregnant or breastfeeding participant (evaluated at baseline)
* Participant unable to read and write in Italian language and to autonomously fill in questionnaires and scales (evaluated at enrolment)
* Participants enrolled in any clinical study receiving experimental treatments for PNH (evaluated at baseline)
* Hypersensitivity to the active substance or to any of the excipient of the study drug.
* Participants with unresolved N. meningitidis infection at treatment initiation
* Participants who are not currently vaccinated against N. meningitidis unless they receive prophylactic treatment with appropriate antibiotics until 2 weeks after vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with documented diagnosis of PNH that were already treated with eculizumab and started treatment with ravulizumab and met the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage Change In Lactate Dehydrogenase (LDH) From Baseline To End Of Observation | Baseline through up to Week 52
  The analysis using descriptive statistics will be performed on the Full Analysis Set, including the participants having the LDH evaluation at both the baseline and at the end of observation.

SECONDARY OUTCOMES:
Percentage Change In LDH From Baseline To End Of Observation On Participants Treated With Ravulizumab With Respect To The Observed Treatment Period With Eculizumab | Baseline through up to Week 52
  The difference of percentage change in LDH from baseline to end of observation will be calculated on participants treated with ravulizumab (over the 52 weeks after baseline) and on the same participants treated with eculizumab (during up to 52 weeks before baseline).
Number of Transfusions During Treatment Period With Ravulizumab | Baseline through up to Week 52
  The number of participants who needed transfusions, with relative frequency and percentage, and descriptive statistics on the total number of transfusions (number of packed red blood cell units transfused) will be calculated for both the treatment period with ravulizumab and the treatment period with eculizumab.
Total Number Of Transfusion Sessions During The Treatment Period With Ravulizumab | Baseline through up to Week 52
  The number of participants who needed transfusions, with relative frequency and percentage, and descriptive statistics on the number of transfusion sessions (number of days) will be calculated for both the treatment period with ravulizumab and the treatment period with eculizumab.
Number Of Participants Undergoing Ravulizumab Without A ≥ 2 gram/deciliter (g/dL) Decrease In Hemoglobin Level In The Absence Of Transfusion | Baseline through up to Week 52
  The proportion of participants without a ≥ 2 g/dL decrease in hemoglobin level in the absence of transfusion will be calculated for both the treatment period with ravulizumab and the treatment period with eculizumab.
Breakthrough Hemolysis (BTH) In The Presence Of Elevated LDH During Treatment Period With Ravulizumab | Baseline through up to Week 52
  BTH is defined as at least 1 new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, dyspnea, anemia [hemoglobin < 10 g/dL], major adverse vascular event including thrombosis, dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥ 2 * upper limit of normal (ULN) after prior LDH reduction to < 1.5 * ULN while on therapy.
Change From Baseline To Each Timepoint Of Assessment Using Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale | Baseline through up to Week 52
  The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Participants will score each item on a 5-point scale. Total scores range from 0 to 52, with a higher score indicating better Quality of Life (QoL).
Change From Baseline To Each Timepoint Of Assessment Using European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 Scale | Baseline through up to Week 52
  EORTC is a questionnaire developed to assess the QoL of cancer participants over the preceding 7 days. The questionnaire has 30 questions related to QoL, with the first 28 questions scored on a 4-point scale and the final 2 questions that probe the participant's overall health and QoL scored on a scale of 1 (very poor) to 7 (excellent). Each subscale has a range of 0 to 100%. Thus, a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
PNH-specific Patient Preference Questionnaire (PPQ) | Week 52
  PNH-PPQ is a participant-centered approach for evaluating preferences for the treatment of PNH. It contains 11 questions assessing overall treatment preference, evaluating treatment preference according to 9 treatment characteristics, assessing the most important treatment characteristic for participant overall medication preference, and evaluating those same aspects of treatment with ravulizumab.
Number of Participants Experiencing Adverse Events (AEs) | Baseline through up to Week 52
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. AEs that will occur during the ravulizumab treatment will be collected and will be reported to the Investigator or qualified designee by the participant.
Costs Related to PNH Sustained By National Health System (NHS) For Ravulizumab Treatment | Baseline, Weeks 18, 34, and 52
  The following medical costs related to PNH sustained by NHS will be collected: specialist visits, pharmacological and non-pharmacological treatments, hospital and emergency rooms admissions, and examinations (by examination type). This will be reported through descriptive statistics and will be appraised considering the quantity of resource consumption by medical resources and its unit costs.
Costs Sustained By The Participants Related To The Infusion Visits For Ravulizumab Treatment | Baseline, Weeks 18, 34, and 52
  The following costs sustained by the participants related to the infusion visits will be collected: average cost to reach the structure, overall time required for the infusion (time to reach the structure + time of infusion), retirement status of the participant, loss of working days, and need of a caregiver. This will be calculated in terms of the total cost of transport and overall time required for infusion.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Clinical Trial Site, Brescia
  - Clinical Trial Site, Catania
  - Clinical Trial Site, Lecce
  - Clinical Trial Site, Ragusa
  - Clinical Trial Site, Roma
  - Clinical Trial Site, Salerno

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Iori AP, De Vivo A, Di Bona E, Caocci G, Fioritoni F, Ciceri F, Beggiato E, Rapezzi D, Amendola A, Figuera A, Selleri C, Longu F, Fattizzo B, Tucci A, Cignetti A, Amico V, Sica S, Metafuni E, Raso S, Urbano TA, Marano L, Di Renzo N, Spedini P, Rambaldi A, Lanza F, Clissa C, Danesin C, Greve MB, Cabibbo S, Ori A, Cassanelli F, Sottana F, Campolo B, Gasparri G, Carini F, Barcellini W. Real life use of ravulizumab in Italian patients with paroxysmal nocturnal hemoglobinuria: evidence from the REACTION observational study. Ann Hematol. 2026 Jan 22;105(2):50. doi: 10.1007/s00277-026-06792-w. PMID 41566054